CLINICAL TRIAL: NCT00229099
Title: A Randomized, Multi-Center, Open Label Trial to Establish the Therapeutic Equivalence Between GerEpo and Eprex® and to Determine the Long Term Safety Profile of GerEpo in Patients on Hemodialysis.
Brief Title: Efficacy and Safety Study of GerEPO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ministry of Health, Malaysia (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT05-02
Record Dates: First submitted 2005-09-28; First posted 2005-09-29 (Estimated); Last update posted 2006-10-26 (Estimated); Status verified 2005-12

CONDITIONS: Chronic Renal Failure Related Anemia

INTERVENTIONS:
Drug: GerEPO

SUMMARY:
The purpose of the study is to establish the equivalence of GerEpo with the standard treatment Eprex® for a treatment period of 12 weeks in patients on Hemodialysis with respect to hemoglobin response and to establish the longer-term safety profile of GerEpo, with special regards for the occurrence of Pure Red Cell Aplasia (PRCA) and other immunogenicity related adverse event

DETAILED DESCRIPTION:
270 patients on Hemodialysis from 25 participating sites who meet inclusion/exclusion criteria will be enrolled into the trial. At the end of the comparative trial, subjects on either arm of the study may opt to enter a longer term cohort study designed to establish the longer-term safety profile of GerEpo, with special regards for the occurrence of Pure Red Cell Aplasia (PRCA) and other immunogenicity related adverse event.

This second part of the study is also opened to all subjects who have given written informed consent, and have ESRF with CRF related anemia who according to current guideline should be treated with Epoetin. Subjects need not be included in the first part of the study.

All patients shall be treated with GerEpo and thereafter observed for at least 1 year to actively monitor for the occurrence of PRCA and other immunogenicity related adverse events. The cohort study shall continue until at least 10,000 patient-years of observation have accrued on the study database.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained.
2. Patients age between 18 and 70 years.
3. Patients who are medically stable on hemodialysis for a minimum of 3 months.
4. Patients on Eprex® treatment for CRF related anemia and maintaining Hb level at or above 9 g/dL(90g/L) while on a stable dose (no change in dose) of Epoetin within 6 weeks preceding the screening phase of this study.
5. Patients who have a serum ferritin level greater than 100μg/L and/or transferrin saturation at least 20% within 3 months preceding the screening phase of this study.

Exclusion Criteria:

1. Pregnant or nursing woman, or women of childbearing potential without an effective method of birth control. Effective birth control methods are oral contraception, Norplant, surgical sterilization, IUD or diaphragms in conjunction with spermicidal foam and condom on the male partner.
2. Participation in any drug trial in which the patient received an Epoetin investigational drug within 30 days preceding the screening phase of this study.
3. Those persons directly involved in the conduct of the study.
4. Poorly controlled hypertension with diastolic blood pressures persistently greater than 110 mmHg at baseline observation.
5. History of seizure disorder.
6. Active acute or chronic infection or inflammatory disease.
7. Any illness that had required hospitalization within the last one month.
8. Had blood transfusion within the last three months.
9. Significant hematologic abnormalities (Evidence of hemolysis by laboratory tests, unexplained acquired microcytosis, thrombocytosis (>500,000/mm3))
10. Severe hyperparathyroidism
11. Diagnosed to have malignant tumor or who have residual tumor after anti-cancer therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270
Dates: Start 2005-04; Study Completion 2005-11

PRIMARY OUTCOMES:
To establish the therapeutic equivalence of GerEpo with the standard treatment Eprex® for a treatment period of 12 weeks in patients on Hemodialysis with respect to hemoglobin response.

SECONDARY OUTCOMES:
• To compare GerEpo with Eprex® with respect to their respective frequency of adverse events
To monitor the occurrence of PRCA and other immunogenicity related adverse events among patients on GerEpo observed for at least a year on therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Zaki Morad, MRCP, FRCP, Principal Investigator — Ministry of Health
Locations (32):
- Malaysia (32):
  - Hospital Sultanah Aminah, Johor Bharu, Johor
  - Pontian Rotary Haemodialysis Centre, Pontian Besar, Johor
  - Hospital Alor Setar, Alor Star, Kedah
  - Hospital Kota Bharu, Kota Bharu, Kelantan
  - SP Menon Dialysis Centre, Kuala Lumpur, Kuala Lumpur
  - Pusat Hemodialisis, Yayasan Felda, Kuala Lumpur, Kuala Lumpur
  - The Kidney Dialysis Centre, Kuala Lumpur, Kuala Lumpur
  - Pantai Medical Centre, Kuala Lumpur, Kuala Lumpur, Kuala Lumpur
  - Hospital Kuala Lumpur, Kuala Lumpur, Kuala Lumpur
  - Tung Shin Hospital, Kuala Lumpur, Kuala Lumpur
  - Hospital Melaka, Malacca, Melaka
  - Pusat Hemodialisis Mawar (Seremban), Seremban, Negeri Sembilan
  - Seremban General Hospital, Seremban, Negeri Sembilan
  - Hospital Tengku Ampuan Afzan, Kuantan, Pahang
  - Pahang Buddhist Association, Kuantan, Pahang
  - Hospital Ipoh, Ipoh, Perak
  - Hospital Taiping, Taiping, Perak
  - Hospital Kangar, Kangar, Perlis
  - Asia Renal Care,Bukit Mertajam, Bukit Mertajam, Pulau Pinang
  - Penang General Hospital, Pulau Pinang, Pulau Pinang
  - Persatuan Buah Pinggang Sabah, Kota Kinabalu, Sabah
  - Hospital Queen Elizabeth, Kota Kinabalu, Sabah
  - Timberland Medical Centre, Kuching, Sarawak
  - MAA Medicare Kidney Charity Dialysis Centre, Kuching, Sarawak
  - Hospital Umum Sarawak, Kuching, Sarawak
  - Ampang Putri Specialist Hospital, Ampang, Selangor
  - Hospital Selayang, Batu Caves, Selangor
  - Hospital Tengku Ampuan Rahimah, Klang, Selangor
  - SP Menon Dialysis Centre, Klang, Selangor
  - Haemodialysis Unit , Sunway Medical Centre, Petaling Jaya, Selangor
  - SP Menon Dialysis Centre, Megah Medical Specialist Centre, Petaling Jaya, Selangor
  - Hospital Kuala Terengganu, Kuala Terengganu, Terengganu

REFERENCES:
- [Derived] Chung EY, Palmer SC, Saglimbene VM, Craig JC, Tonelli M, Strippoli GF. Erythropoiesis-stimulating agents for anaemia in adults with chronic kidney disease: a network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 13;2(2):CD010590. doi: 10.1002/14651858.CD010590.pub3. PMID 36791280
- [Derived] Goh BL, Ong LM, Sivanandam S, Lim TO, Morad Z; Biogeneric EPO Study Group. Randomized trial on the therapeutic equivalence between Eprex and GerEPO in patients on haemodialysis. Nephrology (Carlton). 2007 Oct;12(5):431-6. doi: 10.1111/j.1440-1797.2007.00831.x. PMID 17803464
- See also: the link is an academic research organisation for the trial — http://www.crc.gov.my